CLINICAL TRIAL: NCT01435005
Title: Breast Cancer and Exercise Trial in Alberta: The BETA Trial
Brief Title: Breast Cancer and Exercise Trial in Alberta
Acronym: BETA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Principal Investigator, Christine Friedenreich, Dr. Christine Friedenreich - Study Principal Investigator, AHS Cancer Control Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACF:24404
Record Dates: First submitted 2011-08-30; First posted 2011-09-15 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Breast Neoplasms
Keywords: Prevention and control; Exercise; Sedentary lifestyle; Biological markers
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Sedentary Behavior | interventions — Hospitals, High-Volume

STUDY DESIGN:
Intervention Model Description: Phase 3 - To compare the effects of a high versus moderate volume exercise intervention on specific biological intermediate endpoints for breast cancer in a group of previously inactive postmenopausal women.
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Volume (Active Comparator): Participate in one year of high volume (300 minutes per week) aerobic exercise with free provision of a personal trainer, membership to an exercise facility, body composition assessment.
  Interventions: Other: High Volume
- Moderate Volume (Active Comparator): Participate in one year of moderate volume (150 minutes per week) aerobic exercise with free provision of a personal trainer, membership to an exercise facility, body composition assessment.
  Interventions: Other: Moderate Volume

INTERVENTIONS:
Other: Moderate Volume — Moderate volume (150 minutes per week) aerobic exercise
  Arms: Moderate Volume
Other: High Volume — Participate in one-year high volume (300 minutes per week)aerobic exercise.
  Arms: High Volume

SUMMARY:
The Breast Cancer and Exercise Trial (BETA Trial) is a randomized controlled trial aimed at understanding what dose (or volume) of exercise will best reduce the risk for breast cancer, particularly among women who are between the ages of 50-74. The primary aim is to compare the effects of a high versus moderate volume exercise intervention on specific biological intermediate endpoints for breast cancer in a group of previously inactive postmenopausal women

DETAILED DESCRIPTION:
Overview The proposed project is an evolution from a previous randomized controlled intervention trial conducted by the applicants known as the Alberta Physical Activity and Breast Cancer Prevention (ALPHA) Trial that examined how a one-year aerobic exercise intervention, as compared to a usual sedentary lifestyle, influenced specific hypothesized biologic mechanisms in the association between physical activity and breast cancer risk. In the proposed project, we plan to extend this research to examine how a one-year high versus moderate volume aerobic exercise intervention influences established and novel biologic mechanisms thought to influence breast cancer risk. We are specifically interested in studying what dose of exercise is required to influence the biologic mechanisms involved in breast cancer etiology.

Rationale and Significance Inadequate physical activity, high total caloric intake, and obesity, central adiposity and weight gain throughout lifetime are all clearly associated with increased postmenopausal breast cancer risk and are some of the few risk factors amenable to intervention. Over one third of breast cancer can be attributed to these three risk factors. The exact dose and type of physical activity required for breast cancer risk reduction, however, are unknown. No trials have been conducted that have systematically examined how different volumes of activity influence mechanisms in breast cancer etiology.

Study Aims The primary aim is to compare the effects of a high versus moderate volume exercise intervention on specific hormonal and biological intermediate endpoints for breast cancer in a group of previously sedentary postmenopausal women. The primary objectives will examine the effects of the interventions on measures of adiposity, insulin resistance, sex hormone levels, markers of obesity and inflammation and serum vitamin D. The secondary aim is to evaluate the impact of the high versus moderate exercise interventions among postmenopausal, sedentary women on psychosocial factors. The secondary objectives will compare the effects of the exercise interventions on quality of life and perceived stress among the participants. Adherence to the exercise intervention at 12 and maintenance of exercise at 24 months will also be assessed.

Research Plan A two-centered, two-armed randomized controlled trial is proposed. In total, 330 postmenopausal, sedentary women aged 50-74 years will be recruited from the screening programs and through media campaigns. Strict eligibility criteria will be applied to ensure that women enrolled in the study can be expected to have a change in breast cancer risk over the one-year long intervention. Randomization will be stratified on centre (Calgary or Edmonton) and on body mass index (< or ≥27.5). The intervention arm will undertake aerobic exercise sessions of 300 mins/week for 12 months. The control arm will be asked to undertake 150 mins/week for 12 months. Baseline and 12-month measurements of adiposity (done by computerized tomography and dual energy X-ray absorbitometry scans), fitness, diet, physical activity, quality of life and stress, determinants of exercise adherence and medical, health and demographic characteristics will be made. Bloods, drawn at baseline, six and 12 months, will be assayed to measure estrone, estradiol, testosterone, androstenedione, insulin, glucose, adiponectin, leptin, interleukin-6, tumour necrosing factor-alpha, C-reactive protein and serum hydroxyvitamin D. One year after completion of the study, maintenance of physical and dietary habits will be measured. Intent-to-treat analysis will be used with a Laird-Ware mixed effects model to compare the changes from the baseline to 12-month follow-up. These data will be of direct relevance for effectiveness trials of exercise and diet for breast cancer prevention and for refinement of physical activity guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50- 74 years, postmenopausal women
* No previous cancer diagnosis
* Physically fit to undertake exercise program
* Pass the Physical Activity Readiness
* Medical Exam,acceptable heart and lung function during a sub-maximal treadmill test
* Body mass index : 22 - 40
* Non-users of exogenous hormones or drugs related to estrogen metabolism, breast tissue growth
* Non-Smoker and non-excessive alcohol drinkers
* Residents of Calgary and Edmonton able to attend fitness facility regularly.

Exclusion Criteria:

* < 50 years of age
* Diabetes
* Deemed too fit or too unfit on sub-maximal treadmill test
* Non English Speaking
* > 4 consecutive weeks absence during the intervention period

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Body Fat | 36 Months
  Body composition (including weight, hip circumference, waist circumference, waist-hip ratio, total body fat, subcutaneous fat, intra-abdominal fat, lean body mass, body mass index)

SECONDARY OUTCOMES:
Insulin resistance | 36 months
  Measurements taken of Insulin Levels, Glucose Levels, Insulin Resistance (HOMA Score)
Sex Hormone Levels | 36 months
  Measure levels of Estrone, Estradiol, Androstenedione and Testosterone
Inflammation | 36 months
  Measure levels of C-Reactive protein, Interleukin-6 and Tumour necrosis factor.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Friedenreich, PhD, Principal Investigator — Tom Baker Cancer Centre
Locations (2):
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Centre, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalo-Encabo P, McNeil J, Perez-Lopez A, Valades D, Courneya KS, Friedenreich CM. Weight Regain and Breast Cancer-Related Biomarkers Following an Exercise Intervention in Postmenopausal Women. Cancer Epidemiol Biomarkers Prev. 2021 Jun;30(6):1260-1269. doi: 10.1158/1055-9965.EPI-20-1652. Epub 2021 Mar 18. PMID 33737300
- [Derived] Brenner DR, Ruan Y, Adams SC, Courneya KS, Friedenreich CM. The impact of exercise on growth factors (VEGF and FGF2): results from a 12-month randomized intervention trial. Eur Rev Aging Phys Act. 2019 Jun 24;16:8. doi: 10.1186/s11556-019-0215-4. eCollection 2019. PMID 31285780
- [Derived] Friedenreich CM, Ruan Y, Duha A, Courneya KS. Exercise Dose Effects on Body Fat 12 Months after an Exercise Intervention: Follow-up from a Randomized Controlled Trial. J Obes. 2019 Jan 20;2019:3916416. doi: 10.1155/2019/3916416. eCollection 2019. PMID 30805213
- [Derived] Stone CR, Friedenreich CM, O'Reilly R, Farris MS, Vallerand JR, Kang DW, Courneya KS. Predictors of Adherence to Different Volumes of Exercise in the Breast Cancer and Exercise Trial in Alberta. Ann Behav Med. 2019 Mar 28;53(5):453-465. doi: 10.1093/abm/kay057. PMID 30020401
- [Derived] McNeil J, Farris MS, Ruan Y, Merry H, Lynch BM, Matthews CE, Courneya KS, Friedenreich CM. Effects of prescribed aerobic exercise volume on physical activity and sedentary time in postmenopausal women: a randomized controlled trial. Int J Behav Nutr Phys Act. 2018 Mar 21;15(1):27. doi: 10.1186/s12966-018-0659-3. PMID 29562927
- [Derived] Brenner DR, Ruan Y, Morielli AR, Courneya KS, Friedenreich CM. Physical activity does not alter prolactin levels in post-menopausal women: results from a dose-response randomized controlled trial. Eur Rev Aging Phys Act. 2017 Jul 13;14:10. doi: 10.1186/s11556-017-0179-1. eCollection 2017. PMID 28717404
- [Derived] McNeil J, Brenner DR, Courneya KS, Friedenreich CM. Dose-response effects of aerobic exercise on energy compensation in postmenopausal women: combined results from two randomized controlled trials. Int J Obes (Lond). 2017 Aug;41(8):1196-1202. doi: 10.1038/ijo.2017.87. Epub 2017 Mar 31. PMID 28360432
- [Derived] Courneya KS, McNeil J, O'Reilly R, Morielli AR, Friedenreich CM. Dose-Response Effects of Aerobic Exercise on Quality of Life in Postmenopausal Women: Results from the Breast Cancer and Exercise Trial in Alberta (BETA). Ann Behav Med. 2017 Jun;51(3):356-364. doi: 10.1007/s12160-016-9859-8. PMID 27837524
- [Derived] Friedenreich CM, Neilson HK, Wang Q, Stanczyk FZ, Yasui Y, Duha A, MacLaughlin S, Kallal C, Forbes CC, Courneya KS. Effects of exercise dose on endogenous estrogens in postmenopausal women: a randomized trial. Endocr Relat Cancer. 2015 Oct;22(5):863-76. doi: 10.1530/ERC-15-0243. PMID 26338699
- [Derived] Friedenreich CM, Neilson HK, O'Reilly R, Duha A, Yasui Y, Morielli AR, Adams SC, Courneya KS. Effects of a High vs Moderate Volume of Aerobic Exercise on Adiposity Outcomes in Postmenopausal Women: A Randomized Clinical Trial. JAMA Oncol. 2015 Sep;1(6):766-76. doi: 10.1001/jamaoncol.2015.2239. PMID 26181634
- [Derived] Friedenreich CM, MacLaughlin S, Neilson HK, Stanczyk FZ, Yasui Y, Duha A, Lynch BM, Kallal C, Courneya KS. Study design and methods for the Breast Cancer and Exercise Trial in Alberta (BETA). BMC Cancer. 2014 Dec 6;14:919. doi: 10.1186/1471-2407-14-919. PMID 25480020